CLINICAL TRIAL: NCT03945773
Title: A Phase II, Multicentre, Open-label Study of Cabozantinib as 2nd Line Treatment in Subjects With Unresectable, Locally Advanced or Metastatic Renal Cell Carcinoma With a Clear-Cell Component Who Progressed After 1st Line Treatment With Checkpoint Inhibitors.
Brief Title: Study of Cabozantinib as 2nd Line Treatment in Subjects With Locally Advanced or Metastatic Renal Cell Carcinoma (RCC) With a Clear-Cell Component Who Progressed After 1st Line Treatment With Checkpoint Inhibitors
Acronym: CaboPoint
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F-FR-60000-023; 2018-002820-18 (EudraCT Number)
Record Dates: First submitted 2019-05-09; First posted 2019-05-10 (Actual); Results first posted 2024-12-19 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced or Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort A (Experimental): Subjects who radiographically progressed after one prior line by CPI therapy with ipilimumab and nivolumab.
  Interventions: Drug: Cabozantinib
- Cohort B (Experimental): Subjects who radiographically progressed after one prior line by CPI therapy combined with VEGF-targeted therapy.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — Oral tablets of 60mg, 40mg and 20 mg.
  Other Names: Cabometyx

SUMMARY:
The overall objective of this study is to evaluate the efficacy and safety of cabozantinib as 2nd line treatment in subjects with unresectable, locally advanced or metastatic RCC with a clear-cell component, who progressed after prior Checkpoint Inhibitors (CPI) therapy with ipilimumab and nivolumab in combination or CPI combined with Vascular Endothelial Growth Factor (VEGF)-targeted therapy.

ELIGIBILITY:
Inclusion Criteria:

All subjects must fulfil all the following criteria to be included in the study:

1. Subjects must provide a signed informed consent prior to any study-related procedures;
2. Male or female subjects must be aged ≥18 years on the day the informed consent is signed;
3. Subjects must have histologically confirmed unresectable, locally advanced (defined as disease not eligible for curative surgery or radiation therapy) or metastatic RCC with a clear-cell carcinoma component;
4. Subjects must have radiographic disease progression, according to Investigator's judgement following 1st line treatment with CPI (ipilimumab plus nivolumab) (Cohort A) or CPI in combination with VEGF-targeted therapy (Cohort B);
5. Subjects present ≥1 target lesion according to RECIST 1.1 per Investigator;
6. Subjects should have Eastern Cooperative Oncology Group (ECOG) status 0-1;
7. Subjects with treated brain metastases are eligible if metastases have been shown to be stable as per Investigator's judgement;
8. Subjects must have adequate organ and marrow function, based upon meeting all of the following laboratory criteria within 15 days before baseline:

   1. Absolute neutrophil count (ANC) ≥ 1500/mm3 (≥ 1.5 GI/L).
   2. Platelets ≥ 100,000/mm3 (≥ 100 GI/L).
   3. Haemoglobin ≥ 9 g/dL (≥ 90 g/L).
   4. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 3.0 × upper limit of normal (ULN).
   5. Total bilirubin ≤ 1.5 × ULN. For subjects with Gilbert's disease ≤ 3 mg/dL (≤ 51.3 μmol/L).
   6. Serum creatinine ≤ 2.0 × ULN or calculated creatinine clearance ≥ 30 mL/min (≥ 0.5 mL/sec) using the Cockcroft-Gault equation
   7. Urine protein-to-creatinine ratio (UPCR) ≤ 1 mg/mg (≤ 113.2 mg/mmol) creatinine or 24-hour urine protein < 1 g.
9. Subject must have recovered to baseline or ≤ Grade 1 per CTCAE v5 from toxicities related to any prior treatments, unless Adverse Events (AE(s)) are clinically nonsignificant and/or stable on supportive therapy as determined by the Investigator;
10. Subject must have completed a steroid taper if he/she had an immune-related adverse event associated with immune CPI;
11. Female subjects of childbearing potential (i.e. less than or equal to 2 years postmenopause and not surgically sterile) must provide a negative pregnancy test within 7 days prior to the start of study treatment. If a urine test cannot be confirmed as negative, a negative serum pregnancy test is required;
12. Female subjects of childbearing potential (i.e. less than or equal to 2 years post-menopause and not surgically sterile) and their partners must agree to use highly effective methods of contraception that alone or in combination result in a failure rate of less than 1% per year when used consistently and correctly during the course of the study and for 4 months after the last dose of study treatment;
13. All male participants must agree to refrain from donating sperm and unprotected sexual intercourse with female partners during the study and for 120 days after the last dose of study treatment;
14. Subjects must be willing and able to comply with study requirements, remain at the investigational site for the required duration of each study visit and be willing to return to the investigational site for the follow up evaluation, as specified in the protocol
15. Subjects must be covered by social security or be the beneficiary of such a system (only applicable for French subjects).

Exclusion Criteria:

Subjects will not be included in the study if the subject:

1. Inability to swallow tablets;
2. Was treated with any other investigational medicinal product (IMP) within the last 30 days before baseline;
3. Was previously treated with cabozantinib;
4. Has a contraindication to Magnetic Resonance Imaging (MRI) or contrast medium used for Contrast Tomography (CT)-scan;
5. Presents untreated brain or leptomeningeal metastases, or current clinical or radiographic progression of known brain metastases;
6. Has a diagnosis of a serious cardiovascular disorder:

   1. Congestive heart failure New York Heart Association class 3 or 4, unstable angina pectoris, or serious cardiac arrhythmias;
   2. Uncontrolled hypertension, defined as sustained blood pressure (BP) (>140 mm Hg systolic or >90 mm Hg diastolic pressure) despite optimal antihypertensive treatment;
   3. Stroke (including transient ischaemic attack (TIA)), myocardial infarction (MI) or other ischaemic event, or thromboembolic event (e.g. deep venous thrombosis, pulmonary embolism) within 6 months before screening;
   4. History of risk factors for torsades de pointes (e.g., long QT syndrome);
7. Is receiving concomitant anticoagulation with coumarin agents (e.g. warfarin), direct thrombin inhibitor dabigatran, Direct Factor Xa inhibitors betrixaban or platelet inhibitors (e.g. clopidogrel); Note: The following are allowed anticoagulants: prophylactic use of low-dose aspirin for cardioprotection (per local applicable guidelines) and low dose, low molecular weight heparin (LMWH) are permitted. Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in patients without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before baseline without clinically significant hemorrhagic complications from the anticoagulation regimen or the tumour.
8. Has a gastrointestinal (GI) disorder including those associated with a high risk of perforation or fistula formation:

   (a) Tumours invading the GI tract, active peptic ulcer disease, inflammatory bowel disease, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis or acute obstruction of the pancreatic or biliary duct, or gastric outlet obstruction; b) Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before screening; Note: Complete healing of an intra-abdominal abscess must have been confirmed before screening
9. Presents a corrected QT (QTc) interval calculated by the Fridericia formula (QTcF) > 500 msec within 1 month prior to baseline; Note: If a single ECG shows a QTcF with an absolute value > 500 ms, two additional ECGs at intervals of approximately 3 min must be performed within 30 min after the initial ECG, and the average of these three consecutive results for QTcF will be used to determine eligibility
10. Presents clinically significant haematuria, hematemesis, or haemoptysis of >0.5 teaspoon (2.5 mL) of red blood, or other history of significant bleeding (e.g.

    pulmonary haemorrhage) within 3 months before screening;
11. Presents cavitating pulmonary lesion(s) or known endobronchial disease manifestation;
12. Presents lesions invading major pulmonary blood vessels;
13. Has been diagnosed with other clinically significant disorders such as:

    1. Serious nonhealing wound/ulcer/bone fracture;
    2. Malabsorption syndrome;
    3. Uncompensated/symptomatic hypothyroidism;
    4. Moderate to severe hepatic impairment (Child-Pugh B or C);
    5. Requirement for haemodialysis or peritoneal dialysis;
    6. History of solid organ transplantation;
14. Has a predicted life expectancy of less than 3 months;
15. Has had prior surgery within 4 weeks prior to baseline. Note: If the subject has undergone major surgery, complete wound healing must have occurred 1 month prior to baseline
16. Has had palliative radiation therapy for bone within 2 weeks or for radiation fields including viscera within 4 weeks prior to baseline. Note: Resolution/healing of side effects must be complete prior to baseline;
17. Has a history of another active malignancy within 3 years from screening except for locally curable cancers that have been apparently cured, such as low-grade thyroid carcinoma, prostate cancer not requiring treatment (Gleason Grade ≤6), basal or squamous cell skin cancer, superficial bladder cancer, in situ melanoma, in situ prostate, cervix or breast carcinoma or other treated malignancies with <5% chance of relapse according to the Investigator;
18. Has a history of allergy to study treatment components or agents with a similar chemical structure or any excipient used in the formulation as listed in the Summary of Product Characteristics (SmPC) document;
19. Has rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption are also excluded;
20. Has a serious medical or psychiatric condition that renders the subject unable to understand the nature, scope and possible consequences of the study, and/or presents an uncooperative attitude;
21. Is pregnant or breastfeeding. A β-human chorionic gonadotrophin (HCG) serum pregnancy test will be performed up to 7 days prior to baseline for all female subjects of childbearing potential (i.e. less than or equal to 2 years post-menopause and not surgically sterile);
22. Is likely to require treatment during the study with drugs that are not permitted by the study protocol;
23. Has abnormal baseline findings, any other medical condition(s) or laboratory findings that, in the opinion of the Investigator, might jeopardise the subject's safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2030-12-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (40):
- SALK - Salzburger Landesklinik, Salzburg, Austria
- France (12):
  - CHRU Besançon, Besançon
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Institut de Cancérologie de Lorraine, Nancy
  - CHU de Nîmes - Institut de Cancérologie du Gard, Nîmes
  - Institut Mutualiste Montsouris, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - CHU Strasbourg, Strasbourg
  - Institut Claudius Régaud, Toulouse
  - Gustave Roussy, Villejuif
- Germany (11):
  - Universitätsmedzin Charité, Berlin
  - University Hospital Carl Gustav Carus Dresden, Dresden
  - Universitätsklinikum Essen, Essen
  - University Cancer Center Hamburg Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Klinikum Der Friedrich-Schiller-Universitaet Jena, Jena
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Otto-von-Guericke-Universität University hospital Magdeburg, Magdeburg
  - University, Hospital Münster, Münster
  - Caritas Krankenhaus St.Josef Klinik für Urologie, Regensburg
  - University Hospital Tuebingen, Tübingen
- Netherlands (4):
  - The Netherlands Cancer Institute - Oncology, Amsterdam
  - Maxima Medisch Centrum, Eindhoven
  - Leiden University Medical Center, Leiden
  - Universitair Medisch Centrum Utrecht, Utrecht
- Spain (4):
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Hospital Lucus Augusti, Lugo
  - M.D. Anderson Center Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Switzerland (3):
  - Universitätsspital Bern, Inselspital, Bern
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital St. Gallen, Sankt Gallen
- United Kingdom (5):
  - Western General Hospital - Edinburgh Cancer Centre, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasgow
  - The Christie NHS Foundation Trust, Manchester
  - Mount Vernon Hospital, Northwood
  - Royal Cornwall Hospital (RCH) - Sunrise Centre, Truro

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and/or EU.
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/

REFERENCES:
- [Derived] Albiges L, Schmidinger M, Taguieva-Pioger N, Perol D, Grunwald V, Guemas E. CaboPoint: a phase II study of cabozantinib as second-line treatment in patients with metastatic renal cell carcinoma. Future Oncol. 2022 Mar;18(8):915-926. doi: 10.2217/fon-2021-1006. Epub 2021 Dec 16. PMID 34911359
- See also: Lay language results summary — https://www.ipsen.com/websites/ipsen_com_v2/wp-content/uploads/2025/01/29153832/F-FR-60000-023-Lay-Results-Summary-1.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase II, open-label study was conducted in participants with unresectable, locally advanced or metastatic renal cell carcinoma with a clear-cell component who progressed after 1st line treatment with checkpoint inhibitors (CPI) at 40 sites in 7 countries (Austria, France, Germany, Netherlands, Spain, Switzerland, and the United Kingdom). First participant was recruited on 08 January 2020 and data cut-off (DCO) date was 13 November 2023.
Pre-assignment Details: The study consisted of screening period (within 15 days prior to first cabozantinib dose), treatment period (up to end of study {EOS} [18 months after last participant included in study started cabozantinib treatment]), and post-treatment follow-up period (until participant expired/EOS, whichever occurred first). Participants who continued to benefit from treatment at EOS entered Treatment Extension Phase. A total of 127 participants enrolled. Results are presented up to DCO of 13 November 2023.
Groups:
- Cohort A: Participants who had radiographically progressed after 1 prior treatment with CPI therapy combined with ipilimumab and nivolumab received cabozantinib 60 milligrams (mg) orally once daily (q.d.) until end of the study, disease progression, unacceptable toxicity or withdrawal of consent.
- Cohort B: Participants who had radiographically progressed after 1 prior treatment with CPI therapy combined with vascular endothelial growth factor (VEGF)-targeted therapy received cabozantinib 60 mg orally q.d. until end of the study, disease progression, unacceptable toxicity or withdrawal of consent.
Period: Overall Study
Arm/Group | Cohort A | Cohort B
Started | 85 | 42
Completed | 31 | 16
Not Completed | 54 | 26
Not completed — Consent Withdrawn | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 46 | 22
Not completed — Physician Decision | 1 | 0
Not completed — Other | 1 | 0
Not completed — Ongoing at the time of DCO | 4 | 3

BASELINE CHARACTERISTICS:
Population: Safety population included all included participants who received at least 1 dose of study medication.
Groups:
- Cohort A: Participants who had radiographically progressed after 1 prior treatment with CPI therapy combined with ipilimumab and nivolumab received cabozantinib 60 mg orally q.d. until end of the study, disease progression, unacceptable toxicity or withdrawal of consent.
- Cohort B: Participants who had radiographically progressed after 1 prior treatment with CPI therapy combined with VEGF-targeted therapy received cabozantinib 60 mg orally q.d. until end of the study, disease progression, unacceptable toxicity or withdrawal of consent.
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 85 | 42 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (9.0) | 66.2 (9.7) | 64.2 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 9 | 31
  Male | 63 | 33 | 96
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 50 | 35 | 85
  Missing | 35 | 7 | 42

OUTCOME MEASURES:

1. Primary Outcome: Cohort A: Objective Response Rate (ORR) Assessed by Independent Central Review
Description: ORR was defined as the percentage of participants who achieved a partial response (PR) or complete response (CR) at any timepoint as determined by independent central review per Response Evaluation Criteria in Solid Tumours (RECIST) 1.1. The CR was defined as disappearance of all target lesions. The PR was defined as at least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. The confidence interval of the ORR was calculated using Clopper-Pearson exact method.
Time Frame: Tumour assessments performed at Screening/Baseline (within 28 days prior start of study treatment) and every 12 weeks, up to approximately 40 months
Population: The Efficacy population - Independent Radiology Committee (IRC) included all participants who received at least 1 dose of study medication and provided a baseline assessment for the tumour according to RECIST 1.1, i.e. reported at least 1 target lesion at baseline based on IRC assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A
Number analyzed (Participants) | 79
percentage of participants | 40.5 [29.6 to 52.1]

2. Secondary Outcome: Time to Response (TTR) Assessed by Independent Central Review and Investigator
Description: TTR was defined as the time from start of study treatment to the date of first evidence of response (PR or CR as determined by independent central review and Investigator per RECIST 1.1). The CR was defined as disappearance of all target lesions. The PR was defined as at least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR.
Time Frame: as for outcome 1
Population: Efficacy population-IRC=participants who received at least 1 dose of study medication; provided baseline assessment for tumour per RECIST 1.1, i.e. reported at least 1 target lesion at baseline per IRC assessment. Efficacy population-Investigator=participants who received at least 1 dose of study medication; provided baseline assessment for tumour per RECIST 1.1, i.e. reported at least 1 target lesion at baseline per Investigator assessment. Only participants with response are analyzed.
Measure: Median (Full Range); unit: months
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 42 | 14
months
  Independent Central Review Assessment: number analyzed (Participants) | 32 | 11
  Independent Central Review Assessment | 2.8 [2.4 to 13.8] | 2.8 [2.7 to 8.3]
  Investigator Assessment | 2.8 [1.8 to 19.1] | 2.8 [2.5 to 22.1]

3. Secondary Outcome: Duration of Response (DOR) Assessed by Independent Central Review and Investigator
Description: DOR was defined as the time from first documented response (PR or CR as determined by independent central review and Investigator per RECIST 1.1) to either disease progression (as determined by independent central review and Investigator per RECIST 1.1) or death due to any cause, whichever occurs first. The CR was defined as disappearance of all target lesions. The PR was defined as at least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. The progressive disease (PD) was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters at prior timepoints (including baseline). In addition to the relative increase of 20%, the sum of diameters must also demonstrate an absolute increase of ≥ 5 millimeters (mm). DOR was calculated using the Kaplan-Meier method.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 42 | 14
months
  Independent Central Review Assessment: number analyzed (Participants) | 32 | 11
  Independent Central Review Assessment | NA [11.6 to NA] — NA indicates that the median and upper limit of 95% confidence interval (CI) were not estimable due to insufficient number of participants with events. | 8.3 [5.6 to NA] — NA indicates that the upper limit of 95% CI was not estimable due to insufficient number of participants with events.
  Investigator Assessment | 11.2 [8.3 to 16.7] | 8.3 [3.7 to 11.1]

4. Secondary Outcome: Disease Control Rate (DCR) Assessed by Independent Central Review and Investigator
Description: DCR was defined as the percentage of participants who achieved a PR, CR or stable disease (SD) as determined by independent central review and Investigator per RECIST 1.1. The CR was defined as disappearance of all target lesions. The PR was defined as at least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. The SD was defined as neither sufficient shrinkage to qualify for CR or PR nor sufficient increase to qualify for PD. The PD was defined at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters at prior timepoints (including baseline). In addition to the relative increase of 20%, the sum of diameters must also demonstrate an absolute increase of ≥ 5 mm.
Time Frame: as for outcome 1
Population: Efficacy population-IRC=all participants who received at least 1 dose of study medication and provided baseline assessment for tumour according to RECIST 1.1, i.e. reported at least 1 target lesion at baseline based on IRC assessment. Efficacy population-Investigator=all participants who received at least 1 dose of study medication and provided baseline assessment for tumour according to RECIST 1.1, i.e. reported at least 1 target lesion at baseline based on Investigator assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 85 | 42
percentage of participants
  Independent Central Review Assessment: number analyzed (Participants) | 79 | 40
  Independent Central Review Assessment | 84.8 [75.0 to 91.9] | 82.5 [67.2 to 92.7]
  Investigator Assessment | 83.5 [73.9 to 90.7] | 81.0 [65.9 to 91.4]

5. Secondary Outcome: Progression-free Survival (PFS) Assessed by Independent Central Review and Investigator
Description: PFS was defined as the time from start of study treatment to either disease progression (as determined by independent central review and Investigator per RECIST 1.1) or death due to any cause, whichever occurs first. The PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters at prior timepoints (including baseline). In addition to the relative increase of 20%, the sum of diameters must also demonstrate an absolute increase of ≥ 5 mm. PFS was calculated using the Kaplan-Meier method.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 85 | 42
months
  Independent Central Review Assessment: number analyzed (Participants) | 79 | 40
  Independent Central Review Assessment | 10.9 [8.2 to 14.2] | 8.3 [5.6 to 11.1]
  Investigator Assessment | 10.9 [8.2 to 13.6] | 8.2 [5.6 to 9.2]

6. Secondary Outcome: Cohort B: Objective Response Rate Assessed by Independent Central Review
Description: ORR was defined as the percentage of participants who achieved a PR or CR at any timepoint as determined by independent central review per RECIST 1.1. The CR was defined as disappearance of all target lesions. The PR was defined as at least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. The CI of the ORR was calculated using Clopper-Pearson exact method.
Time Frame: as for outcome 1
Population: The Efficacy population - IRC included all participants who received at least 1 dose of study medication and provided a baseline assessment for the tumour according to RECIST 1.1, i.e. reported at least 1 target lesion at baseline based on IRC assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort B
Number analyzed (Participants) | 40
percentage of participants | 27.5 [14.6 to 43.9]

7. Secondary Outcome: Objective Response Rate Assessed by Investigator
Description: ORR was defined as the percentage of participants who achieved a PR or CR at any timepoint as determined by Investigator per RECIST 1.1. The CR was defined as disappearance of all target lesions. The PR was defined as at least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. The CI of the ORR was calculated using Clopper-Pearson exact method.
Time Frame: as for outcome 1
Population: The Efficacy population - Investigator included all participants who received at least 1 dose of study medication and provided a baseline assessment for the tumour according to RECIST 1.1, i.e. reported at least 1 target lesion at baseline based on Investigator assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 85 | 42
percentage of participants | 49.4 [38.4 to 60.5] | 33.3 [19.6 to 49.5]

8. Secondary Outcome: Overall Survival (OS) Assessed by Investigator
Description: OS was defined as the time from the start of treatment until death due to any cause. OS was calculated using the Kaplan-Meier method.
Time Frame: From the start of study treatment (Day 1) up to end of study, 45 months
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 85 | 42
months | 24.3 [18.5 to 31.8] | 24.1 [17.1 to NA] — NA indicates that the upper limit of 95% CI was not estimable due to insufficient number of participants with events.

9. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Kidney Cancer Symptom Index (FKSI-DRS) Score at Month 40
Description: The FKSI-DRS questionnaire consisted of 9-items to evaluate participant's symptoms in the past 7 days such as lack of energy, pain, weight-loss, bone-pain, shortness of breath, fatigue, fever, blood in urine etc. Participants rated each question from 0 (not at all) to 4 (very much). Total score was calculated as the sum of the item responses divided by the number of items completed and multiplied by the total number of items in the scale. Total score ranged from 0 to 36. Higher scores indicated less symptoms. Baseline was defined as the last questionnaire answered prior to the first dose of study drug. A negative change from baseline indicated worse outcome.
Time Frame: Baseline (Day 1) and Month 40
Population: The Efficacy population - Investigator included all participants who received at least 1 dose of study medication and provided a baseline assessment for the tumour according to RECIST 1.1, i.e. reported at least 1 target lesion at baseline based on Investigator assessment. Only participants with data collected at Baseline and Month 40 are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 37 | 22
score on a scale | -3.0 (5.4) | -2.4 (5.6)

ADVERSE EVENTS:
Time Frame: TEAEs are reported from first dose of study treatment (Day 1) up to 30 days post last dose of study treatment, 46 months. Results are presented up to DCO of 13 November 2023.
Description: The safety population included all participants who received at least 1 dose of study medication.
Arm/Group | Cohort A | Cohort B
All-Cause Mortality (participants affected / at risk) | 46/85 | 22/42
Serious Adverse Events (participants affected / at risk) | 51/85 | 15/42
Other Adverse Events (participants affected / at risk) | 85/85 | 41/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=85) | Cohort B (N=42)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 2 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 1 (2)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diaphragmatic hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Femoral hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Jejunal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis necrotising (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 8 (8) | 5 (5)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Abdominal wall wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Radicular pain (Nervous system disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=85) | Cohort B (N=42)
Anaemia (Blood and lymphatic system disorders) | 9 (9) | 6 (7)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Hypothyroidism (Endocrine disorders) | 25 (26) | 13 (13)
Diarrhoea (Gastrointestinal disorders) | 60 (99) | 31 (54)
Stomatitis (Gastrointestinal disorders) | 33 (45) | 20 (26)
Nausea (Gastrointestinal disorders) | 27 (33) | 12 (14)
Constipation (Gastrointestinal disorders) | 23 (30) | 10 (11)
Vomiting (Gastrointestinal disorders) | 15 (18) | 10 (14)
Abdominal pain (Gastrointestinal disorders) | 13 (14) | 4 (6)
Haemorrhoids (Gastrointestinal disorders) | 9 (10) | 4 (6)
Dry mouth (Gastrointestinal disorders) | 7 (8) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 8 (9) | 1 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 (8) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 3 (3)
Oral dysaesthesia (Gastrointestinal disorders) | 5 (5) | 1 (1)
Toothache (Gastrointestinal disorders) | 6 (6) | 0 (0)
Fatigue (General disorders) | 32 (45) | 19 (22)
Asthenia (General disorders) | 23 (34) | 6 (9)
Oedema peripheral (General disorders) | 6 (7) | 4 (6)
Mucosal inflammation (General disorders) | 7 (8) | 2 (3)
Pyrexia (General disorders) | 7 (8) | 0 (0)
Chest pain (General disorders) | 1 (1) | 3 (4)
Hepatic cytolysis (Hepatobiliary disorders) | 9 (11) | 1 (1)
Urinary tract infection (Infections and infestations) | 9 (12) | 4 (5)
Nasopharyngitis (Infections and infestations) | 5 (9) | 2 (3)
Oral candidiasis (Infections and infestations) | 5 (5) | 0 (0)
Alanine aminotransferase increased (Investigations) | 19 (22) | 13 (16)
Aspartate aminotransferase increased (Investigations) | 18 (24) | 14 (15)
Weight decreased (Investigations) | 16 (16) | 6 (7)
Blood thyroid stimulating hormone increased (Investigations) | 5 (5) | 8 (12)
Blood alkaline phosphatase increased (Investigations) | 8 (8) | 2 (2)
Blood creatinine increased (Investigations) | 5 (5) | 4 (5)
Gamma-glutamyltransferase increased (Investigations) | 7 (7) | 2 (2)
Blood bilirubin increased (Investigations) | 5 (6) | 3 (5)
Platelet count decreased (Investigations) | 4 (5) | 3 (3)
Blood lactate dehydrogenase increased (Investigations) | 2 (2) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 41 (51) | 23 (25)
Hypocalcaemia (Metabolism and nutrition disorders) | 5 (7) | 11 (14)
Hypophosphataemia (Metabolism and nutrition disorders) | 7 (13) | 5 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 9 (9) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (12) | 3 (6)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 (4) | 4 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5 (6) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 17 (21) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (14) | 7 (10)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (8) | 8 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (11) | 6 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (9) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Dysgeusia (Nervous system disorders) | 20 (25) | 5 (5)
Headache (Nervous system disorders) | 10 (11) | 6 (7)
Dizziness (Nervous system disorders) | 12 (13) | 1 (2)
Ageusia (Nervous system disorders) | 1 (1) | 3 (3)
Lethargy (Nervous system disorders) | 1 (1) | 3 (5)
Proteinuria (Renal and urinary disorders) | 13 (16) | 6 (8)
Haematuria (Renal and urinary disorders) | 3 (4) | 4 (6)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 18 (19) | 8 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 (19) | 8 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (14) | 8 (9)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 39 (50) | 10 (20)
Dry skin (Skin and subcutaneous tissue disorders) | 10 (10) | 10 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (13) | 8 (10)
Rash (Skin and subcutaneous tissue disorders) | 11 (19) | 4 (7)
Hair colour changes (Skin and subcutaneous tissue disorders) | 8 (8) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (4)
Hypertension (Vascular disorders) | 43 (56) | 20 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-02-23): https://cdn.clinicaltrials.gov/large-docs/73/NCT03945773/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-17): https://cdn.clinicaltrials.gov/large-docs/73/NCT03945773/SAP_001.pdf